



Official Title: The Effect of Cognition Targeted Physical Therapy in People With Non-

specific Neck Pain: A Mixed-Method Multiple Case Study

**Project:** Physical Therapy in people with Neck Pain

ID: HR01\_MCS\_NeckPain

**NCT ID:** Not yet assigned

**Date of document:** 1-11-2021





## INFORMED CONSENT FORM PARTICIPANTS

Project: Physical Therapy in People with Neck Pain

- I have read and understood the information about the project, as provided in the information letter. I have been given the opportunity to ask questions about the project and I had enough time to decide about my participation. My questions have been answered sufficiently.
- I understand that taking part in this research project is voluntarily. I understand that I can end my participation at any time without giving reasons.
- I understand that other researchers will have access to this data. These researchers are mentioned in the information letter.
- I give permission for the collection and use of my data for the purposes stated in the information letter.
- I give permission to store my data at the research location for another 15 years after this research project.
- I hereby give my permission to contact me after this research for a follow-up research:
  - o Yes
  - o No
- I want to be informed about the general results of this study:
  - o Yes
  - o No
- I want to participate to this research project

| Name Participant: | |
|---|---|
| Signature: | Date:/ |
| I declare that I have fully informed this participant re<br>Name researcher: | egarding this research project. |
| Signature: | Date:// |